CLINICAL TRIAL: NCT03924934
Title: Community-associated Highly-Resistant Enterobacterales
Acronym: COCARE
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-3017; 1R01AI143910 (NIH)
Record Dates: First submitted 2019-04-03; First posted 2019-04-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Enterobacteriaceae Infections; Community-Acquired Infections; Healthcare Associated Infection; Carbapenem-Resistant Enterobacteriaceae Infection
Keywords: Infection; Bacterial Infection; CRE; Enterobacterales
MeSH Terms: conditions — Enterobacteriaceae Infections; Community-Acquired Infections; Cross Infection; Infections; Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — HRE that are recovered either from clinical samples or from Biowipe samples will be sent to a central research laboratory for species confirmation and antibacterial susceptibility testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Possible CA-HRE: Patients with suspected CA-HRE, discharged home after a previous hospitalization or outpatient visit during which CA-HRE was isolated from a clinical culture (approximately 210 patients)
- HA-HRE: Hospitalized patients with healthcare-associated HRE, who are not discharged home (HA-HRE) (210 selected control patients)
- HA-HRE discharged home: Patients eventually discharged home, either directly or through another facility, after a hospitalization during which HA-HRE was isolated from a clinical culture (100)
- Community contacts: Contacts of patients with HRE (approximately 1,500)

SUMMARY:
This is a prospective multi-center study. Bacterial isolates from hospitalized patients with CA-HRE will be compared to those from hospitalized patients with healthcare-associated HRE (HA-HRE). In addition, community spread of CRE will be determined.

DETAILED DESCRIPTION:
Patients who are discharged home from the hospital and meet criteria for possible CA-HRE will be recruited. These index participants will be interviewed to determine the epidemiologic network, and will be mailed a monthly BioWipe kit to screen for ongoing HRE intestinal carriage. Contacts of the index participant will also be approached and mailed a BioWipe kit to screen for the presence of HRE and/or carbapenemase gene(s) that were present in the index patient. If this initial sample is negative, the contact is not further interviewed or tested. If the initial screening is positive for the carbapenemase gene of interest, then the contact will be asked to answer the same questions as the index patient and will receive a monthly BioWipe kit. For each positive contact, a second-generation network of contacts will be constructed, who in turn will be approached for screening.

An additional subset of participants, those with CDC-defined HRE isolated during hospitalization who are not discharged home will also be included. All HRE isolates that are isolated from the patient as part of routine clinical care will be sub-cultured and shipped to the central research laboratory. A limited data set will be collected.

ELIGIBILITY:
Inclusion Criteria:

Category 1: Patients who live at home and meet the following criteria:

* CDC-defined HRE isolated during a previous hospitalization or outpatient visit
* Home origin
* First positive HRE culture within 48 hours of admission (in case of hospitalization)

Category 2: Hospitalized patients with CDC-defined HRE isolated during hospitalization who are not discharged home and who meet any of the following criteria:

* Admitted from other care facility (not home origin)
* Do not have first positive HRE culture within 48 hours of admission

Category 3: Patients with CDC-defined HRE isolated during a previous hospitalization or outpatient visit who are eventually discharged home and who meet any of the following criteria:

* Admitted from other care facility (not home origin)
* Do not have first positive HRE culture within 48 hours of admission (in case of hospitalization)

Category 4: Participants who meet the following criteria:

• Community contact of a participant in Category 1 and/or 3.

Exclusion Criteria:

In all categories, participants who meet the following criteria will be excluded:

• Age <18 years

In category 1, the following are exclusionary:

* pre-existing renal failure
* pre-existing liver disease
* immunocompromised
* history of malignancy
* pregnancy

In addition, in category 1, 3 and 4, who meet the following criteria will be excluded:

• Unable to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four categories of participants will be included:
  1. Patients with suspected CA-HRE, discharged home after a previous hospitalization or outpatient visit during which CA-HRE was isolated from a clinical culture (approximately 210 patients)
  2. Hospitalized patients with healthcare-associated HRE, who are not discharged home (HA-HRE) (210 selected control patients)
  3. Patients eventually discharged home either directly or through another facility after a hospitalization or outpatient visit during which HA-HRE was isolated from a clinical culture (100)
  4. Contacts of patients with HRE (approximately 1,500)
Sampling Method: Non-Probability Sample
Enrollment: 2172 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of CA-HRE infections | enrollment - end of study, up to approximately 1 year
  Proportion of HRE cases diagnosed in hospitalized patients that are community-associated out of all CRE cases in hospitalized patients
Proportion of HRE-culture positive community contacts of hospitalized patients with HRE as determined by stool culture. | enrollment - end of study, up to approximately 1 year
  In community contacts of patients discharged from the hospital after HRE diagnosis, the presence or absence of HRE in stool samples will be determined by culture. Then, the total number of community contacts with HRE-positive stool cultures will be divided by the total number of tested community contacts to derive the proportion of community contacts with stool cultures positive for HRE.

CONTACTS AND LOCATIONS:
Overall Officials: David van Duin, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9-36 months following publication
Access Criteria: IRB approval, DUA executed